CLINICAL TRIAL: NCT00062309
Title: A Phase III Intensity Modulated Radiotherapy Dose Escalation Trial for Prostate Cancer Using Hypofractionation
Brief Title: Comparison of Two Radiation Therapy Regimens in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304712; P30CA006927 (NIH); FCCC-02602
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: stage II prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIMRT (Active Comparator): 76 Gy in 38 fractions
  Interventions: Radiation: radiation therapy
- HIMRT (Experimental): 70.2 Gy in 26 fractions
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays and other sources of radiation to kill tumor cells. It is not yet known which radiation therapy regimen is more effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is comparing two different regimens of radiation therapy to see how well they work in treating patients with stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of conventional intensity-modulated radiotherapy (IMRT) vs hypofractionated IMRT, in terms of freedom from biochemical failure in men with intermediate- to high-risk prostate cancer.
* Compare the local control, freedom from distant metastasis, and overall survival of patients treated with these regimens.
* Determine local failure, using biopsy of the prostate, when objective tests (prostate-specific antigen, ultrasound, and digital rectal exam) suggest relapse in these patients.
* Compare the extent of disease eradication using biopsy of the prostate at 2 years after therapy in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the impact of these regimens on patient preferences and utilities.

OUTLINE: This is a randomized study. Patients are stratified according to pretreatment prostate-specific antigen (no greater than 10 ng/mL vs greater than 10 to 20 ng/mL vs greater than 20 ng/mL), Gleason score (5-7 vs 8-10), and risk status (high risk vs intermediate risk). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo conventional intensity-modulated radiotherapy (IMRT) 5 days a week for 7.5 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo hypofractionated IMRT 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity.

Patients with high-risk disease also undergo androgen deprivation therapy for 2 years.

Quality of life is assessed at baseline, every 6 months for 1 year, and then annually for 4 years.

Patients are followed at 3 months, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinical stage T1b-T3c disease
  * No clinical or radiographic evidence of metastasis
* Prostate-specific antigen (PSA) less than 80 ng/mL
* Gleason score at least 5
* One of the following criteria must be met:

  * PSA greater than 10 ng/mL
  * Gleason score greater than 6
  * T2b or greater palpable disease
  * Three or more biopsy cores involved with a Gleason score of at least 5

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other medical condition that would preclude study participation
* No other active malignancy within the past 5 years except nonmetastatic skin cancer or early stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic leukemia)
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No more than 4 months of prior androgen deprivation therapy
* Neoadjuvant and adjuvant androgen deprivation therapy is allowed for high-risk disease only

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* No prior or planned radical prostate surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2002-06; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Freedom from biochemical and/or disease failure rates | weekly during treatment, at 3 months, 6 months or 2 years then yearly

CONTACTS AND LOCATIONS:
Overall Officials: Mark Buyyounouski, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Pollack A, Bae K, Khor LY, et al.: Stability of tumor biomarkers in archival tissue from men treated with radiotherapy for prostate cancer: an analysis of RTOG 92-02 and Fox Chase randomized trials. [Abstract] Int J Biol Markers 22 (1): 72-3, 2006.
- [Derived] Avkshtol V, Ruth KJ, Ross EA, Hallman MA, Greenberg RE, Price RA Jr, Leachman B, Uzzo RG, Ma C, Chen D, Geynisman DM, Sobczak ML, Zhang E, Wong JK, Pollack A, Horwitz EM. Ten-Year Update of a Randomized, Prospective Trial of Conventional Fractionated Versus Moderate Hypofractionated Radiation Therapy for Localized Prostate Cancer. J Clin Oncol. 2020 May 20;38(15):1676-1684. doi: 10.1200/JCO.19.01485. Epub 2020 Mar 2. PMID 32119599
- [Derived] Pollack A, Walker G, Horwitz EM, Price R, Feigenberg S, Konski AA, Stoyanova R, Movsas B, Greenberg RE, Uzzo RG, Ma C, Buyyounouski MK. Randomized trial of hypofractionated external-beam radiotherapy for prostate cancer. J Clin Oncol. 2013 Nov 1;31(31):3860-8. doi: 10.1200/JCO.2013.51.1972. Epub 2013 Oct 7. PMID 24101042